CLINICAL TRIAL: NCT01112228
Title: Assessing Clinical Staging Tools for Tracking the Impacts of Obesity on Individuals
Brief Title: Clinical Staging Tools for the Impacts of Obesity on Individuals
Acronym: COST
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: Clinical Obesity Staging Tools
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Results first posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obese patients: Obese patients for Bariatric surgery
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — Bariatric surgery: Gastric bypass, Sleeve gastrectomy, or Gastric banding

SUMMARY:
This study will assess various published staging tools to assess the health impacts of obesity on individuals. The aim is to identify benefits and drawbacks, and thus help Obesity Centres and GPs better assess obese individuals as well as better identify who benefits most from having weight loss treatment.

DETAILED DESCRIPTION:
This study will assess various published staging tools to assess the health impacts of obesity on individuals. The aim is to identify benefits and drawbacks, and thus help Obesity Centres and GPs better assess obese individuals as well as better identify who benefits most from having weight loss treatment

ELIGIBILITY:
Inclusion Criteria:

* Morbid obesity
* At least 1 year follow-up after bariatric surgery

Exclusion Criteria:

* N/A

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with BMI > 40 or >35 and a obesity-related medical condition
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2009-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carek le Roux, MD PhD, Study Chair — Imperial College London
Locations (1):
- Imperial Weight Centre, Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aasheim ET, Aylwin SJ, Radhakrishnan ST, Sood AS, Jovanovic A, Olbers T, le Roux CW. Assessment of obesity beyond body mass index to determine benefit of treatment. Clin Obes. 2011 Apr;1(2-3):77-84. doi: 10.1111/j.1758-8111.2011.00017.x. Epub 2011 Jul 5. PMID 25585572

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Obese Patients
Started | 600
Completed | 600
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Obese Patients
Number analyzed (Participants) | 600
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 48 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 420
  Male | 180
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 600
  Unknown or Not Reported | 0
BMI (kg/m2 ) [Mean (Standard Deviation); unit: kg/m^2] | 49 (12)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Obesity Scores After Weight Loss Treatment
Description: Changes were measured in the following clinical domains
  -Airway, Body Mass Index, Cardiovascular risk, Diabetes, Economic, Functional. Gonadal, Body Image.
  An improvement was considered when any 1 of these domains changes for the positive. Thus, if a patient had an improvement in cardiovascular risk the intervention was considered beneficial even if no other domains changed.
  Out measure is calculated as the count of participants achieving at least 1 improvement (Count)
Time Frame: Minimum of 1 year follow-up
Population: Obese patients for Bariatric surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Obese Patients
Number analyzed (Participants) | 600
Participants | 600

2. Secondary Outcome: Changes in Obesity Scores in Various Subgroups
Description: Changes in obesity scores in patients with carious co-morbid conditions (eg, type 2 diabetes, sleep apnoea) before bariatric surgery
Time Frame: Minimum of 1 year follow-up
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Diabetes and Obesity: Patients with diabetes pre-surgery who had improvement in any one of the clinical domains as measure in the King's Obesity Staging Score
- Patients With Sleep Apnea: Patients with Sleep Apnea pre-surgery who had improvement in any one of the clinical domains as measured in the King's Obesity Staging Score
Arm/Group | Patients With Diabetes and Obesity | Patients With Sleep Apnea
Number analyzed (Participants) | 130 | 96
Participants | 130 | 96

ADVERSE EVENTS:
Time Frame: 1 year
Description: As per usual
Arm/Group | Obese Patients
All-Cause Mortality (participants affected / at risk) | 0/600
Serious Adverse Events (participants affected / at risk) | 0/600
Other Adverse Events (participants affected / at risk) | 30/600
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obese Patients (N=600)
Abdominal pain (Gastrointestinal disorders) | 30 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes